CLINICAL TRIAL: NCT01518283
Title: Phase II Study of Weekly Cabazitaxel for Advanced Prostate Cancer in "Unfit" Hormone-Refractory Patients Previously Treated With Docetaxel
Brief Title: Study of Weekly Cabazitaxel for Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABASEM-SOGUG
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2015-11

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: Weekly cabazitaxel.; Advanced Hormone-refractory prostate Cancer.; Unfit patients.
MeSH Terms: interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel (Experimental): Drug: Cabazitaxel 10 mg/m2
  Interventions: Drug: Cabazitaxel 10 mg/m2

INTERVENTIONS:
Drug: Cabazitaxel 10 mg/m2 — Cabazitaxel 10 mg/m2 in a 1-hour infusion on days 1, 8, 15 and 22 of 5-week cycles.
  Other Names: Jevtana

SUMMARY:
This is a multicenter open label non randomized phase II clinical trial of Weekly Cabazitaxel for Advanced Prostate Cancer in Hormone-Refractory Patients Previously Treated with Docetaxel.

The purpose of this study is to evaluate the activity of the weekly administration of cabazitaxel as time to progression by PSA at week 12.

DETAILED DESCRIPTION:
The efficacy of three-weekly cabazitaxel is accompanied by an appreciable rate of serious side effects and toxic deaths. The toxicity rates observed, including grade III-IV neutropenia, febrile neutropenia and diarrhea, could be an obstacle to the use and management of a drug that, on the other hand, has demonstrated great activity. In the treatment of patients with prostate cancer, who have a larger number of morbidities than patients with breast cancer, we assume the risk that in the transition from clinical trial to clinical practice the drug will not be used much because of the risk of side effects, cost, the discomfort derived from the routine use of G-CSF and the lack of patient compliance with this type of regimens.

Rates of neuropathy, nail and conjunctive toxicity with this new taxane are not relevant, which suggests that weekly administration will not produce relevant toxicity problems. Weekly administration of other taxanes improved hematologic tolerance along with a better therapeutic range in some cases, increasing the dose intensity and activity without increasing the associated toxicity.

Phase I study has been reported studying weekly administration of cabazitaxel, recommended dose is 10 mg/m2, administered on days 1, 8, 15 and 22 every 5 weeks in a 1-hour infusion, being diarrhea the dose-limiting toxicity observed in this study.

Given the pharmacokinetic characteristics of this taxane and its activity and toxicity profile, cabazitaxel might be a good candidate for studying in a weekly administration regimen in patients with prostate cancer with a greater risk of toxicity associated with treatment every 3 weeks, such as patients who have received previous pelvic radiation therapy that affects more than 25% of the bone marrow reserve, patients over 75 years with a worse performance status (ECOG 2) or who have already experienced important hematologic toxicity in the previous treatment with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have given written informed consent.
2. Age ≥ 18 years.
3. ECOG 0-2.
4. Patients with a histologic or cytologic diagnosis of advanced prostate cancer (any Gleason grade).
5. Previous and ongoing castration by orchiectomy or LHRH agonists. Antiandrogen must be discontinued prior to study start.
6. Disease progression, clinically or radiologically documented, during or after treatment with docetaxel, with a minimum cumulative dose of 225 mg/m2.
7. "Unfit" patients defined as patients who satisfy at least one of the following criteria:

   * ECOG 2
   * Dose reduction due to febrile neutropenia during the previous treatment with docetaxel
   * Radiation therapy affecting more than 25% of bone marrow reserve
8. Documented metastatic disease and progressing after docetaxel treatment. Progression criteria is considered any of the following three or more than one at once:

   * Progressive elevation of PSA measured in three successive determinations one week difference between them at least;
   * Should be considered progression of measurable disease by RECIST criteria;
   * Bone progression as evidenced by the appearance of two or more new lesions on bone scan.
9. Patients who have received a maximum of one prior chemotherapy for metastatic disease.
10. Prior anticancer therapy should have been interrupted 28 days before the start of study treatment (the patient may have continued treatment with prednisone 5 mg bid.
11. Adequate blood, liver and kidney function:

    * Hemoglobin > 9.0 g/dl
    * ANC > 1.5 x 10*9/L
    * Platelets > 100 x 10*9/L
    * AST/SGOT and ALT/SGPT < 2.5 x ULN
    * Bilirubin < 1.0 x ULN
    * Creatinine <1.5 mg/dL x ULN. If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance <60 mL/min should be excluded (see Annex 7 for formula)
12. Adequate baseline cardiac function (LVEF ≥ 50%).
13. Life expectancy ≥ 12 weeks.
14. Patients must agree to use an effective contraceptive method during treatment with the study drug and up to 1 month after ending the treatment.

Exclusion Criteria:

1. Patients who received radiation therapy that exceeded 40% of the bone marrow reserve or that ended within the last 3 weeks prior to inclusion.
2. If being treated with radiation therapy, should be completed before the three weeks prior to initiation of treatment research.
3. Previous treatment with two or more chemotherapy regimens for metastatic disease. A new line of treatment is also when a patient receives again docetaxel after clinical, radiological or PSA progression to a prior regimen with docetaxel.
4. Previous treatment with chemotherapy or surgery in the last 4 weeks.
5. Peripheral neuropathy or stomatitis ≥ 2 (National Cancer Institute Common Terminology Criteria - NCI CTCAE vs. 4.03).
6. Any other type of cancer in the last 5 years, except for basal cell skin carcinoma.
7. Cerebral or leptomeningeal metastasis.
8. Myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass, congestive heart failure (NYHA class III or IV), stroke or transitory ischemic episodes.
9. Patients who present any severe or uncontrolled medical condition (including uncontrolled diabetes mellitus) or any other condition that may affect the patient's participation and study compliance.
10. Previous treatment with cabazitaxel.
11. Known hypersensitivity (≥ grade 3)to cabazitaxel, polysorbate 80, prednisone or prednisolone, or docetaxel or paclitaxel.
12. Known history of active infection that requires systemic antibiotic or antifungal treatment.
13. Patients who are receiving or expect to receive treatment with strong inhibitors or strong inducers of cytochrome CYP450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments) (see Annexes 5 and 6).
14. Patients being treated with any investigational product.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-05; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Time to progression by PSA at week 12, according to the PCCTWG II criteria. | 12 weeks
  Time to progression by PSA at week 12. PSA progression defined as an increase of ≥25% over nadir PSA concentration provided that the increase in the absolute PSA value was ≥5 μg/L for men with no PSA response, or ≥50% over nadir for PSA responders and PSA responders defined as a reduction in serum PSA concentration of ≥50% in patients with a baseline value of ≥20 μg/L.

SECONDARY OUTCOMES:
time to PSA progression | Patients will be followed until PSA progression, an expected average of 6 months
  Time to PSA progression, according to the PCCTWG II criteria, defined as the time between enrolment and the first date of PSA progression.
biochemical response rate | Patients will be followed until end of treatment, an expected average of 6 months
  Biochemical response by PSA determination defined as the percentage of patients with 30%,50% and 80% reduction respect to baseline in patients with a baseline value >=20 mcg/L confirmed by a repeat PSA measurement after at least 3 weeks.
Objective response rate | Patients will be followed until end of treatment, an expected average of 6 months
  Proportion of patients with an objective tumoral response according to modified RECIST criteria
Overall survival | Patients will be followed until death, an expected average of 18 months
  Overall survival is calculated since the date of patient study enrolment till death.
Evaluate the safety and tolerability profile of cabazitaxel. | 6 months (during treatment)
  All adverse events will be graded according to National Cancer Institute Common Terminology Criteria for adverse events (version 4.03).
  Adverse events, biochemistry, hematology, vital signs and electrocardiograms will be monitored throughout the study.
Pain response | Until end of treatment, an expected average of 6 months
  Determine the pain response in patients with stable pain at baseline by means of the McGill-Melzack MPQ-sf questionnaire, defined as ≥ 2 points with respect to baseline on the PPI scale without increase in the analgesic scale, or with a decrease of ≥ 50% in the use of analgesics without an increase in pain that is maintained for more than 3 weeks.
Correlation between presence-absence of baseline pain with overall survival, time to progression and PSA response rate. | Until death, an expected average of 18 months
Correlation of the Charlson co-morbidity index and ADL/IADL dependency indexes with survival and toxicity | Until death, an expected average of 18 months
Assessment and quantification of Circulating Tumour Cells and level correlation between the beginning of treatment and their variation through treatment with time to progression and overall survival | Until death, an expected average of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Climent, MD, Principal Investigator — FUNDACIÓN INSTITUTO VALENCIANO DE ONCOLOGÍA, Servicio de Oncología Médica, Profesor Beltrán Báguena, 11, 8 y 19, Valencia, 46009
Locations (12):
- Spain (12):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Institut Català D'Oncologia L'Hospitalet (Ico), L'Hospitalet de Llobregat, Barcelona
  - Hospital de Sant Joan de Déu, Manresa, Barcelona
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Hospitalario de Ourense, Ourense
  - Hospital Virgen Del Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia